CLINICAL TRIAL: NCT03852355
Title: the Effectiveness of 3rd Occipital Radiofrequency Versus Systemic Steroid in Headache Management in Rheumatoid Arthritis; a Randomized Controlled Trial
Brief Title: the Effectiveness of 3rd Occipital Radiofrequency Versus Systemic Steroid in Headache Management in Rheumatoid Arthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Emad Zarief , MD, Associate professor, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB17300357
Record Dates: First submitted 2019-02-22; First posted 2019-02-25 (Actual); Last update posted 2020-07-24 (Actual); Status verified 2020-07

CONDITIONS: Rheumatoid Arthritis; Headache
MeSH Terms: conditions — Arthritis, Rheumatoid; Headache | interventions — Steroids

STUDY DESIGN:
Intervention Model Description: To our knowledge the effectiveness of 3rd occipital nerve blocks in managing chronic upper neck pain, headache in RA patients is not measured yet, so we aimed at assessing the the effectiveness of 3rd occipital nerve blocks in headache management in RA patients who used other medical agents and to compare the results with those of the patients who used only 3rd occipital nerve pulsed radiofrequancy on clinical and radiographic bases.
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Radiofrequency (Active Comparator): bilateral 3rd occipital nerve RF under fluoroscopic guidance
  Interventions: Drug: Radiofrequency
- Systemic steroid (Active Comparator): received systemic steroids oral prednisolone tablet, 10 mg/day.
  Interventions: Drug: Steroids

INTERVENTIONS:
Drug: Radiofrequency — ), received bilateral 3rd occipital nerve RF under fluoroscopic guidance. Levobupivacaine (0.3 mL; 0.75%) and triamcilonone (1 mg) were injected at each level
  Arms: Radiofrequency
Drug: Steroids — received systemic steroids oral prednisolone tablet, 10 mg/day
  Arms: Systemic steroid

SUMMARY:
Rheumatoid arthritis is a common type of autoimmune arthritis that is characterized by inflammation of the synovial membranes. Even though any joint can be affected by the disease, cervical spine is often affected, and cervical pain is reported by 40-88% of RA patients, Cervical spine involvement is a feature of long-lasting disease, where atlantoaxial impaction with odontoid process vertical subluxation through the foramen magnum being one of the greatest and dangerous complications

DETAILED DESCRIPTION:
To our knowledge the effectiveness of 3rd occipital nerve blocks in managing chronic upper neck pain, headache in RA patients is not measured yet, so we aimed at assessing the the effectiveness of 3rd occipital nerve blocks in headache management in RA patients who used other medical agents and to compare the results with those of the patients who used only 3rd occipital nerve pulsed radiofrequancy on clinical and radiographic bases.

ELIGIBILITY:
Inclusion Criteria:

* patients suffering from upper neck pain and/or headache due to bilateral 3rd occipital nerve involvement evidenced by magnetic resonance imaging (MRI).

Exclusion Criteria:

* disc herniation with radicular pain,
* symptomatic spinal stenosis,
* surgical interventions of the cervical spine within the last 3 months,
* uncontrolled major depression or psychiatric disorders,
* heavy opioid usage

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2019-02-25 (Actual); Primary Completion 2019-09-10 (Actual); Study Completion 2019-10-25 (Actual)

PRIMARY OUTCOMES:
neck disability index score | 6 months
  maximum score = 50 worst paint , lowest score = no pain

SECONDARY OUTCOMES:
Severity of headache Visual analog scale | 6 months
  maximum scale= 100 worst paint , lowest scale = no pain

CONTACTS AND LOCATIONS:
Locations (1):
- Emad Zarief Kamel Said, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided